CLINICAL TRIAL: NCT03213314
Title: HepaT1ca: Quantifying Liver Health in Surgical Candidates for Liver Malignancies
Acronym: Hepatica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other); Perspectum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AC17009; 223180 (Other: IRAS)
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Liver Cancer; Surgery; Liver Regeneration; Colorectal Cancer Metastatic
Keywords: LiverMultiScan; multiparameter MRI; functional liver remnant; liver resection; hepatic resection; portal vein embolisation; preoperative liver function; postoperative liver failure
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Nested cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Main cohort (Experimental): Patients undergoing liver resection
  Interventions: Diagnostic Test: Multiparameter magnetic resonance imaging
- Nested cohort PVE (Experimental): Patients undergoing liver resection after portal vein embolisation
  Interventions: Diagnostic Test: Multiparameter magnetic resonance imaging
- Nested cohort neoadjuvant chemotherapy (Experimental): Patients undergoing liver resection after neoadjuvant chemotherapy
  Interventions: Diagnostic Test: Multiparameter magnetic resonance imaging
- Nested cohort TACE (Experimental): Patients undergoing trans arterial chemoembolisation for presumed hepatocellular carcinoma
  Interventions: Diagnostic Test: Multiparameter magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Multiparameter magnetic resonance imaging — LiverMultiScan before and after surgery to assess liver health prior to liver resection and in the regenerative phase.
  Other Names: LiverMultiScan

SUMMARY:
This observational clinical cohort study aims to evaluate the clinical utility of LiverMultiScan in quantifying liver health prior to liver resection or TACE. The results will enable further developments in scanning protocols and software, and clearly define the relevance of applying this technology as part of the pre-operative assessment of the patient being considered for liver resection or TACE.

DETAILED DESCRIPTION:
The liver is unique among the abdominal organs for the capacity to regenerate post-operatively. However, a minimum functional liver remnant (FLR) is required for patients to survive the initial perioperative period. At present, the assessment of the FLR is based on volume alone, in the context of clinical judgment and surrogate markers of liver function based on blood tests. Recently, Perspectum Diagnostics have developed and validated LiverMultiScan, an MRI-based technology that can non-invasively quantify fibroinflammatory disease in addition to steatosis and iron content. In this project, we plan to use LiverMultiScan as an additional direct measurement of liver health prior to resectional surgery or transarterial chemoembolization (TACE), so that liver volume and function can be combined. For example, surgery with a predicted FLR of 21% might be survivable if the liver tissue was in extremely good health, whereas surgery with a predicted FLR of 40% might be lethal if the liver tissue was in poor health. Occasionally, portal vein embolization (PVE) is performed to promote hypertrophy of the FLR. Furthermore, non-resectional intervention, for example TACE for primary liver cancers, is well-tolerated by patients with healthy livers, but can lead to serious liver decompensation and liver failure if TACE is delivered to a liver in poor health. Currently, the available imaging modalities are limited in their ability to assess liver health in liver resection or TACE candidates. Liver fat content (steatosis) can be assessed with CT, or more accurately with MRI. However, fibroinflammatory disease, which has been shown to correlate with post-resection morbidity, typically requires an invasive biopsy to diagnose accurately.

This research project will support the definition, development and technical validation of Hepatica, which aims to build on the MRI technology underlying LiverMultiScan and develop the additional functionality required to meet this clinical need.

ELIGIBILITY:
Inclusion Criteria:

* Patients being considered for liver resection

Exclusion Criteria:

* i. Patients under the age of 18 years will be excluded from the present study. ii. Prisoners will be excluded from the present study. iii. Persons unable to have an MRI scan (including but not limited to claustrophobia, implanted metallic devices, metal foreign body) iv. Adults with incapacity v. Non-provision of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Correlation between the pre-operative liver health assessment score and the post-operative liver function composite integer-based risk score. | 24 months
  Correlation between the pre-operative liver health assessment score (Hepatica score - calculated by weighting future remnant liver volume by liver inflammation and fibrosis (LIF) score) and the post-operative liver function composite integer-based risk (Hyder-Pawlik) score.

SECONDARY OUTCOMES:
To compare LiverMultiScan image interpretations with histological findings | 24 months
  To compare LiverMultiScan image interpretations with clinical outcome after surgery in three domains: post-operative liver function, surgery-specific complication rate, and overall complication rate
• To evaluate LiverMultiScan image interpretations correlated with post-operative length of stay. | 24 months
  • To compare LiverMultiScan image interpretations with histological findings in the resected liver specimen in four domains: fibrosis, inflammation, fat content and iron load as title

CONTACTS AND LOCATIONS:
Overall Officials: Damian J Mole, MBChB PhD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Hampshire Hospitals Foundation Trust, Basingstoke
  - NHS Lothian Royal Infirmary of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Controlled access of study data through a reasonable request to the study management team, after a reasonable embargo period after completion of the study

REFERENCES:
- [Derived] Mole DJ, Fallowfield JA, Sherif AE, Kendall T, Semple S, Kelly M, Ridgway G, Connell JJ, McGonigle J, Banerjee R, Brady JM, Zheng X, Hughes M, Neyton L, McClintock J, Tucker G, Nailon H, Patel D, Wackett A, Steven M, Welsh F, Rees M; HepaT1ca Study Group. Quantitative magnetic resonance imaging predicts individual future liver performance after liver resection for cancer. PLoS One. 2020 Dec 2;15(12):e0238568. doi: 10.1371/journal.pone.0238568. eCollection 2020. PMID 33264327
- [Derived] Mole DJ, Fallowfield JA, Kendall TJ, Welsh F, Semple SI, Bachtiar V, Kelly M, Wigmore SJ, James Garden O, Wilman HR, Banerjee R, Rees M, Brady M. Study protocol: HepaT1ca - an observational clinical cohort study to quantify liver health in surgical candidates for liver malignancies. BMC Cancer. 2018 Sep 12;18(1):890. doi: 10.1186/s12885-018-4737-3. PMID 30208871